CLINICAL TRIAL: NCT00852189
Title: A Phase I Study of EC0489 Administered Weeks 1 and 3 of a 4-Week Cycle
Brief Title: Study of EC0489 for the Treatment of Refractory or Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-0489-01
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Cancer
Keywords: Cancer; Phase 1; EC0489; EC20; Refractory; Metastatic; Experimental
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — EC 0489

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EC0489, Injection — PART A: Dose escalation from a starting dose of 1.0 mg/m2 IV bolus on Monday, Wednesday, and Friday Weeks 1 and 3 of a 4-week cycle to the Maximum Tolerated Dose (MTD)
  Other Names: Folic acid desacetylvinblastine hydrazide conjugate
Drug: EC20 — 20-25 mCi 99mTc-EC20 administered IV bolus 1-2 hours prior to imaging and at end of study for subjects who received 1 cycle or more of EC0489.
  Other Names: Folic acid-technetium 99m conjugate; Folatescan
Drug: EC0489, Injection — PART B: Once PART A MTD is determined, PART B will begin. Dose escalation from a starting dose of 4.2 mg/m2 IV bolus once weekly in a 4-week cycle to the Maximum Tolerated Dose (MTD).
  Other Names: Folic acid desacetylvinblastine hydrazide conjugate

SUMMARY:
This is a Phase 1 clinical trial evaluating the safety and tolerability of escalating doses of EC0489 in patients with refractory or metastatic tumors who have exhausted standard therapeutic options.

DETAILED DESCRIPTION:
This is a Phase 1, dose escalation study of EC0489 administered by intravenous bolus (IV) during weeks 1 and 3 of a 4-week cycle in PART A and weekly on a 4-week cycle in PART B.

Both Parts are open to patients with refractory or metastatic cancer who have exhausted standard therapeutic options. EC0489 is a drug that is specifically designed to enter cells via a folate vitamin receptor. Experimental evidence shows that the target receptor is over-expressed in many human cancers. There are no previous human studies of EC0489; however, lab research (research in test tubes or animals) using EC0489 has shown activity against tumors in animals. This activity in animal models suggests that EC0489 may be useful as chemotherapy against human cancers. The primary objective of this study is to determine the safety and maximum tolerated dose of EC0489 given by intravenous bolus. The efficacy of treatment will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histological or cytological diagnosis of neoplasm
* No effective standard therapeutic options
* ECOG performance status of 0-2
* ≥ 4 weeks post therapeutic radiation or recovered (or returned to baseline) from any acute toxicity associated with prior cytotoxic therapy. Patients previously treated with non-cytotoxic therapy (e.g., EGFR, VGEF, etc.) and who have recovered from or have controlled drug-associated toxicity are allowed to enter the trial after a period consisting of 4 half-lives of the agent.
* Negative serum pregnancy test for women of child-bearing potential within one week prior to treatment with investigational agents (99mTc-EC20 and EC0489)and willingness to practice contraceptive methods
* Adequate bone marrow reserve, renal and hepatic function

Exclusion Criteria:

* Concurrent malignancies
* Women who are pregnant or breast-feeding
* Evidence of symptomatic brain metastases
* Receiving concomitant anticancer therapy (excluding supportive care)
* Requires palliative radiotherapy at time of study entry
* Requires antifolate therapy for comorbid conditions
* Heart failure characterized as greater than NYHA Class I
* History of myocardial infarct
* Any of the following baseline echocardiogram findings: valvular lesions (stenosis or insufficiency) characterized as greater than moderate, systolic ventricular impairment characterized as greater than mild, left ventricular ejection fraction < 55%, any feature of the echocardiogram that would confound interpretation of the serial echocardiograms required by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Dose escalation to the highest dose that can be safely administered to produce acceptable, manageable and reversible toxicity in no more than 0 or 1 of 6 patients

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic parameters | Obtained during the first cycle of therapy on Days 1 and 3
Anti-tumor activity | Initial dose of study therapy to disease progression
Uptake of 99mTc-EC20 in tumors and normal tissues | 1-2 hours post administration of 99mTc-EC20
Safety and Tolerability | Initiation of study therapy through 30 day post last dose of study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Messmann, MD, MHS, MSc, Study Director — Endocyte
Locations (6):
- United States (6):
  - Horizon Oncology Center, Lafayette, Indiana
  - Greenebaum Cancer Center - University of Maryland, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute - Wayne State University, Detroit, Michigan
  - Great Lakes Cancer Institute - Michigan State University, Lansing, Michigan
  - Providence Cancer Institute, Southfield, Michigan